CLINICAL TRIAL: NCT05064150
Title: A Cohort Study of Symptom Burden and Therapeutic Selection in Neuroendocrine Tumors (NETs)
Brief Title: Neuroendocrine Tumors - Patient Reported Outcomes
Acronym: NET-PRO
Status: Active, not recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: Allina Health System (Other); Medical College of Wisconsin (Other); University of Kansas Medical Center (Other); University of Texas Southwestern Medical Center (Other); University of Utah (Other); University of Florida (Other); Ohio State University (Other); University of Michigan (Other); University of Pittsburgh Medical Center (Other); Medical University of South Carolina (Other); University of North Carolina, Chapel Hill (Other); Vanderbilt University Medical Center (Other); Mayo Clinic (Other); Northern California CarciNET Community (Unknown); Neuroendocrine Cancer Awareness Network (Unknown); Neuroendocrine Tumor Research Foundation (Unknown); Healing NET Foundation (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Michael A O'Rorke, Assistant Professor, University of Iowa
Other Study IDs: 202104599
Record Dates: First submitted 2021-08-27; First posted 2021-10-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Tumors; Gastroenteropancreatic Neuroendocrine Tumor; Lung Neuroendocrine Neoplasm; Neuroendocrine Carcinoma
Keywords: Patient-reported outcomes; Neuroendocrine; Quality of Life; Survival; Treatment sequencing; Symptom burden
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NET patient observational cohort: Patients diagnosed with lung or gastrointestinal neuroendocrine tumors

SUMMARY:
With so many therapeutic options available (i.e.: biologic therapy, liver directed therapy, radiotherapy and chemotherapy), the purpose of this project is to partner with patients on comparative effectiveness research (CER) to achieve the goal of alleviating undue toxicity, and optimizing effectiveness and sequencing of therapy for neuroendocrine tumors (NET) patients. We will conduct a study of all newly occurring GEP-NET and lung NET cases aged 18 years and older diagnosed between 01/01/2018 through 09/30/2024 across 14 sites participating in the National Patient-Centered Clinical Research Network (PCORnet), enrolling an average of 215 patients per site over the 3 year study period (2515 patients total), allowing up to 60 months of follow-up for medical record outcomes. Participants will complete four online or paper surveys over 18 months; these surveys will focus on patient-reported outcomes, including questions on quality of life, treatment decisions, and experiences with cancer care. Survey data will be linked to participant medical record data to achieve study aims.

DETAILED DESCRIPTION:
NETs are a group of neoplasms that occur most frequently in the gastrointestinal tract, pancreas and the lungs, collectively referred to as gastroenteropancreatic (GEP-NETs) and lung-NETs. There are currently fewer than 180,000 patients living with this condition in the United States, meeting the criteria for rare disease status. NETs are typically slow growing, with vague signs and a myriad of symptoms (carcinoid syndrome) leading to diagnostic delays. Thus, NET patients typically experience a prolonged clinical course with active disease, and many have significant symptom burdens. However, assessment of quality of life outside of therapy trials remains scarce and of poor quality. What's more, over half of GEP-NETs are diagnosed with spread of their disease at diagnosis and are not candidates for curative surgery. Fortunately, many of these tumors are amenable to long-term medical treatment with somatostatin analogues (SSAs)- which slow down the production of hormones, especially serotonin, which helps to control the symptoms of carcinoid syndrome. However, living with distant spread of the disease increases the probability for the disease to progress. Following failure of first-line SSA therapy there are no clear consensus guidelines as to the optimum sequencing of other therapeutic options. NET patients are left wondering not only 'what therapy would be best to try next?', but 'if I were to take this option now, what treatment options will be closed off to me in the future?' and clinicians are unsure as to how best to tailor treatment selection on the characteristics of the patient and their tumor.

There is currently no large nationally recruiting prospective (forward in time) observational study of NET patients. Our large study will robustly generate real-world evidence on the frequency and sequence of commonly used treatments for GEP and lung NET patients in relation to Patient Reported Outcomes (PROs) and survival/progression, endpoints that matter most to NET patients, their caregivers, and clinicians involved in their care. Given the lack of consensus guidelines as to the optimum sequencing of treatments, evidence generated in this study will aid patient (and clinician) navigation and selection of the next most appropriate therapy, accounting for the preferences and needs of the individual patient, whilst respecting the underlying profile of their tumor. Moreover, the infrastructure this study will generate (i.e.: electronic identification of NET patients, entry and completion of tumor table data in PCORnet, and a unique NET patient health record portal), will foster future CER studies in NETs and other rare diseases.

The four specific aims of this project are:

1. To describe the frequency of treatment regimens received by line of therapy, and examine their association with symptom burden and changes in 6, 12 and 18 month health-related quality of life (HRQoL) outcomes. The influence of patient preferences, beliefs, attitudes, and experience of care on choice of these treatment regimens will also be examined.
2. To examine the association of patient, clinical, and tumor characteristics on the selection of first-line and beyond treatment regimens and compare the effects of common treatment sequences on frequency of subsequent treatments received and outcomes of overall survival and disease progression.
3. To compare the effectiveness of peptide receptor radionuclide therapy (PRRT) regimens on outcomes of renal toxicity, disease progression, and patient-reported symptoms and HRQoL.
4. To disseminate lessons learned and expand enrollment of the prospective cohort to patient advocate organizations, and to use the infrastructure developed to aid in the study of other rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adults age 18 years or older at time of NET diagnosis
* (2) Diagnosis of GEP-NET or lung NET between 1/1/2018 and 09/30/2024, as evidenced by
* (a) medical record information on diagnoses and/or medications and/or treatments and/or test results and/or clinical notes and/or procedures and/or encounters and/or tumor characteristics, and
* (b) patient self-attestation of their diagnosis.

Exclusion Criteria:

Any GEP-NET/Lung NET prior to 1/1/18, as evidenced by medical record information on diagnoses and/or medications and/or treatments and/or test results and/or clinical notes and/or procedures and/or encounters and/or tumor characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion/exclusion criteria will be assessed by a combination of a computable phenotype (computer code or algorithm) that is run against participating site electronic medical record and/or tumor registry data holdings, and/or manual review of patient EMR; and patient self-report.
Sampling Method: Non-Probability Sample
Enrollment: 2539 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire (EORTC QLQ-C30) | Change in score across baseline, 6, 12, and 18 month time points.
  Incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. Responses to the QLQ-C30 will be linearly transformed to a 0-100 scale using EORTC guidelines, a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Neuroendocrine Carcinoid Module (EORTC QLQ-GI.NET21) | Change in score across baseline, 6, 12, and 18 month time points.
  The QLQ-GINET21 contains a total of 21 items: four single-item assessments relating to muscle and/or bone pain (MBP), body image (BI), information (INF) and sexual functioning (SX), together with 17 items organized into five proposed scales: endocrine symptoms (ED; three items), GI symptoms (GI; five items), treatment-related symptoms (TR; three items), social functioning (SF) of the new module (SF21; three items) and disease-related worries (DRW; three items). Responses to the QLQ-GINET21 will be linearly transformed to a 0-100 scale using EORTC guidelines, with higher scores reflecting more severe symptoms.
Sequencing of treatment regimens from electronic medical records (% of patients using modality) | Up to 5 years
  Ordering of treatment receipt i.e.: first-line, 2nd line 3rd line therapies
Renal function | Change in score across baseline, 6, 12, and 18 month time points.
  Creatinine clearance loss (per/Yr)

SECONDARY OUTCOMES:
Norfolk Carcinoid Symptom Score | Change in score across baseline, 6, 12, and 18 month time points.
  Patient-reported symptoms
Experiences with cancer care (from CANCORS) | Change in score across baseline, 6, 12, and 18 month time points.
  13 items to assess cancer care as described at https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2953972/
Progression-free survival | 1-, 3-, and 5-year
  Time to event
Overall survival | Up to 5 years
  Time to event
Adverse toxicities | Up to 5 years
  Incident acute renal failure, dialysis and liver failure during follow-up
Presence of Acute Renal Failure Diagnosis | Up to 5 years
  Common Data Model (CDM) diagnosis codes for acute renal failure and dialysis
Health related Quality of Life (HRQoL) by PRRT regimen | Change in score across baseline, 6, 12, and 18 month time points.
  Changes in HRQOL
Symptom scores by PRRT regimen | Change in score across baseline, 6, 12, and 18 month time points.
  Changes in symptom scores
Renal toxicity (creatinine clearance) by PRRT isotope | Up to 5 years
  Creatinine clearance loss (per/Yr) 177Lu vs 90Y
Renal toxicity of PRRT by primary tumor location & grade 3 disease | Up to 5 years
  Creatinine clearance loss (per/Yr) GEP-NETs vs lung NETs and G3

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Rorke, PhD, Principal Investigator — University of Iowa
Locations (14):
- United States (14):
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc, Kansas City, Kansas
  - Regents of the University of Michigan, Ann Arbor, Michigan
  - Allina Health System, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Inc, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to researchers and details will be provided.
Supporting Information: Study Protocol, ICF

DOCUMENTS (1):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT05064150/Prot_000.pdf